CLINICAL TRIAL: NCT02703844
Title: Caloric Vestibular Stimulation in Parkinson's Disease
Brief Title: Vestibular Stimulation in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KENT/DW/PD/2016
Record Dates: First submitted 2016-02-26; First posted 2016-03-09 (Estimated); Results first posted 2022-10-31 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Active (Active Comparator): Participants will be receiving an active Caloric Vestibular Stimulation treatment for a duration of 8 weeks, 7 days a week, twice daily for 19 minutes.
  Interventions: Device: Caloric Vestibular Stimulation
- Placebo (Sham Comparator): Participants will be receiving a Sham Caloric Vestibular Stimulation treatment for a duration of 8 weeks in the same manner as the active arm: 7 days a week, twice daily for 19 minutes.
  Individuals allocated to this arm will be later crossed over, in unblinded fashion, to the active arm if the treatment shows evidence of efficacy and safety.
  Interventions: Device: Sham Caloric Vestibular Stimulation

INTERVENTIONS:
Device: Caloric Vestibular Stimulation — Stimulation of the vestibular nerves
  Arms: Active
Device: Sham Caloric Vestibular Stimulation — Sham stimulation of the vestibular nerves
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether caloric vestibular stimulation improves symptoms of Parkinson's Disease.

DETAILED DESCRIPTION:
Parkinson's Disease (PD) is a nationwide public health problem, inflicting a complex constellation of physical and neuropsychiatric symptoms which are shown to progress with time. This research will investigate the potential of caloric vestibular stimulation (CVS), a non-invasive form of brain stimulation, as a treatment for individuals who suffer from Parkinson's Disease. Investigators will investigate whether core cognitive and physiological deficits are responsive to stimulation by comparing participants' performance on behavioral and physiological measures after baseline and either active or placebo stimulation phases with the aim of drawing initial insights into the application of CVS within this population. The study design is based on a single-case study that recently demonstrated durable, clinically meaningful gains in the motor and nonmotor symptoms of PD.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be diagnosed with idiopathic Parkinson's Disease as defined by the UK PDS Brain Bank Criteria.
* Participants must report limitations to Activities of Daily Life (ADL, UPDRS subscale 2)
* Capacity to consent to the study
* Motivated to comply with the protocol
* An understanding of English sufficient to comply with the protocol
* Spouse/ carer willing to support the participant throughout the study

Exclusion Criteria:

* Diagnosis of induced Parkinson's or essential/dystonic tremor
* Premorbid psychiatric history (including affective disorder, psychosis or deliberate self- harm)
* Previous exposure to neurostimulation
* Inner ear pathology

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2016-03; Primary Completion 2017-10-09 (Actual); Study Completion 2018-07-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Palmer, Study Director — University of Kent (research ethics & governance lead)
Locations (1):
- University of Kent, Canterbury, Kent, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all clinical outcome measures have been made available.
Time Frame: The data is available in an online repository.
Access Criteria: The data is provided in an open-access format.
URL: https://data.mendeley.com/datasets/m7ths6gdv9/1

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants will be receiving a Sham Caloric Vestibular Stimulation treatment for a duration of 8 weeks in the same manner as the active arm: 7 days a week, twice daily for 19 minutes.
  Individuals allocated to this arm will be later crossed over, in unblinded fashion, to the active arm if the treatment shows evidence of efficacy and safety.
  Sham Caloric Vestibular Stimulation: Sham stimulation of the vestibular nerves
Period: Randomized Controlled Portion
Arm/Group | Active | Placebo
Started | 23 | 23
Completed | 16 | 17
Not Completed | 7 | 6
Period: Cross-Over to Active
Arm/Group | Active | Placebo
Started (Cross-over portion was only offered to those who were randomized to placebo in the randomized portion of the study. Not all participants from the placebo group of the randomized controlled period chose to move into the cross-over period and receive active treatment) | 0 | 14
Completed (Participants were allowed to use the active study device for up to 4 months. Completed is those who used the study device for the full 4 months.) | 0 | 5
Not Completed | 0 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active | Placebo | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.7 (11.3) | 72.2 (6.6) | 70.9 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 5 | 16
  Male | 12 | 18 | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Non-Motor Symptom Scale (NMSS) Total Score [Mean (Standard Deviation); unit: score on a scale] | 126.2 (29.8) | 117.7 (32.6) | 122 (31.2)
MDS-UPDRS Part II Score [Mean (Standard Deviation); unit: score on a scale] | 22.5 (9.1) | 21.4 (5.3) | 21.9 (7.4)
MDS-UPDRS Part III Score [Mean (Standard Deviation); unit: score on a scale] | 49.3 (17.6) | 45.4 (16.3) | 47.4 (16.9)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Nonmotor Symptom Severity Scale (NMSS)
Description: The NMSS is a 30-item rater-based scale to assess a wide range of non-motor symptoms in patients with Parkinson's disease (PD). The NMSS measures the severity and frequency of non-motor symptoms across nine dimensions. Score range of 0-360, with 0 being no symptom burden
Time Frame: Change at end of treatment (week 12) relative to the average of two baseline visits
Population: data reported for this outcome includes anyone who received at least one treatment with the study device and had a baseline NMSS performed. Change scores were not normally distributed and therefore nonparametric tests were used and medians are reported
Measure: Median (95% Confidence Interval); unit: change in scale total score
Arm/Group | Active | Placebo
Number analyzed (Participants) | 23 | 23
change in scale total score | -33.5 [-40.3 to -17.7] | -2.0 [-16.5 to 8.3]
Statistical Analysis 1: Comparison: Active vs Placebo; Test type: Superiority; p = 0.0089, ANCOVA

2. Secondary Outcome: Change From Baseline in the MDS-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part II: Motor Aspects of Experiences of Daily Living
Description: The MDS-UPDRS Part II is a 13-item patient-reported assessment of activities of motor aspects of experiences of daily living. Scores range between 0-52, with the higher score indicating greater impairment to activities of daily living
Time Frame: Change at end of treatment (week 12) relative to baseline average
Population: data reported for this outcome includes anyone who received at least one treatment with the study device and had a baseline MDS-UPDRS Part II performed.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Active | Placebo
Number analyzed (Participants) | 23 | 23
score on a scale | -3.2 [-5.1 to -1.2] | -0.4 [-1.7 to 1.0]

3. Secondary Outcome: Change From Baseline in the MDS-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III: Motor Examination
Description: The MDS-UPDRS Part III is a 33-item assessment of motor function evaluated by a trained blinded rater. Scores range between 0-132 with higher scores indicating more severe motor symptoms
Time Frame: Change at end of treatment (week 12) relative to baseline average
Population: data reported for this outcome includes anyone who received at least one treatment with the study device and had a baseline MDS-UPDRS Part III performed.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Active | Placebo
Number analyzed (Participants) | 23 | 23
score on a scale | -8.8 [-12.5 to -5.1] | -2.8 [-7.3 to 1.6]

4. Other Pre Specified Outcome: Change From Baseline in the Montreal Cognitive Assessment
Description: rapid screening instrument for mild cognitive dysfunction, with a score range from zero to 30, with higher being closer to normal
Time Frame: Change at one-month post-treatment follow-up (week 17) relative to baseline average
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Change From Baseline in the Epworth Sleepiness Scale
Description: a brief measure that is commonly used to assess daytime sleepiness in PD and other disorders. Scores can range from 0 to 24. The higher the score, the higher that person's average daytime sleepiness
Time Frame: Change at one-month post-treatment follow-up (week 17) relative to baseline average
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Change From Baseline in the Modified Schwab & England
Description: clinical outcome assessment of an individual's ability to function in activities of daily living
Time Frame: Change at one-month post-treatment follow-up (week 17) relative to baseline average
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Change From Baseline in the 2 Minute Walk
Description: performance measure of walking ability and functional capacity
Time Frame: Change at one-month post-treatment follow-up (week 17) relative to baseline average
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Change From Baseline in the 10 Meter Walk
Description: performance measure used to assess walking speed
Time Frame: Change at one-month post-treatment follow-up (week 17) relative to baseline average
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Change From Baseline in the Timed Up and Go (TUG)
Description: measures gait and the probability of falls in adults
Time Frame: Change at one-month post-treatment follow-up (week 17) relative to baseline average
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Change From Baseline in the Fatigue Severity Scale
Description: questionnaire for evaluating the impact of fatigue. scores range from 9-63 with a higher score for greater fatigue.
Time Frame: Change at one-month post-treatment follow-up (week 17) relative to baseline average
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Change From Baseline in the EuroQol 5D
Description: questionnaire for use in clinical and economic appraisal and population health. scores range from 0-100 for each question with 0 being the worst and 100 being the best
Time Frame: Change at one-month post-treatment follow-up (week 17) relative to baseline average
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Change From Baseline in the SF-12 Health Survey
Description: self-reported outcome measure assessing the impact of health on an individual's everyday life. Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning
Time Frame: Change at one-month post-treatment follow-up (week 17) relative to baseline average
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Change From Baseline in the Hospital Anxiety and Depression Scale
Description: self-rating scale developed to assess psychological distress. scores range between 0-21 with higher scores equaling more severe impairment
Time Frame: Change at one-month post-treatment follow-up (week 17) relative to baseline average
Reporting Status: Not Posted

14. Other Pre Specified Outcome: EEG/Event - Related Potentials Abnormalities - Physiological Measurement
Description: Assessment of any changes to P300 during ERPs and beta wave in a resting state.
Time Frame: Change at end of treatment (week 12) relative to baseline
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 17 weeks
Groups:
- Cross-Over: Participants who received the Sham Caloric Vestibular Stimulation in the Randomized portion of the study will be receiving active caloric Vestibular Stimulation treatment for a duration of up to 4 months, 7 days a week, twice daily for 19 minutes.
  Caloric Vestibular Stimulation: Stimulation of the vestibular nerves
Arm/Group | Active | Placebo | Cross-Over
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23 | 0/14
Serious Adverse Events (participants affected / at risk) | 2/23 | 1/23 | 0/14
Other Adverse Events (participants affected / at risk) | 6/23 | 4/23 | 6/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=23) | Placebo (N=23) | Cross-Over (N=14)
Arm fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | NA
Knee Infection (Infections and infestations) | 1 (1) | 0 (0) | NA
Fainting Episode (Nervous system disorders) | 1 (1) | 0 (0) | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=23) | Placebo (N=23) | Cross-Over (N=14)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0) | 1 (1)
Ear discomfort (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0)
Fall (Nervous system disorders) | 1 (1) | 2 (2) | 4 (4)
Chest Infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-07-25): https://cdn.clinicaltrials.gov/large-docs/44/NCT02703844/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-15): https://cdn.clinicaltrials.gov/large-docs/44/NCT02703844/SAP_001.pdf